CLINICAL TRIAL: NCT03242681
Title: Endoscopy Assisted Probing Versus Simple Probing in Patients With Primary Congenital Nasolacrimal Duct Obstruction: A Randomized Clinical Trial
Brief Title: Endoscopy Assisted Probing Versus Simple Probing in Primary Congenital Nasolacrimal Duct Obstruction
Acronym: Non
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.TUMS.VCR.REC.1395.1200
Record Dates: First submitted 2017-07-23; First posted 2017-08-08 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-03

CONDITIONS: Congenital Nasolacrimal Duct Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopy Assisted Probing (Experimental): Endoscopy Assisted Probing
  Interventions: Procedure: Endoscopy Assisted Probing procedure
- Simple Probing (Active Comparator): Simple Probing
  Interventions: Procedure: Endoscopy Assisted Probing procedure

INTERVENTIONS:
Procedure: Endoscopy Assisted Probing procedure — The patency of the system will be tested by irrigation with 1 ml normal saline. A cannula was introduced via the upper or lower canaliculus as far as the lacrimal sac and fluid injected through the system from a 5 ml syringe. Nasal endoscopy and irrigation will be performed simultaneously and free flow of fluid from the lacrimal sac to the nose will confirm anatomical patency of the system

SUMMARY:
The aim of this study is to compare results of endoscopy assisted nasolacrimal probing with the standard simple probing in cases with congenital nasolacrimal duct obstruction . Furthermore, investigators will identify associated anatomical anomalies. Investigators believe results of this study can be valuable in better understanding of this disease and provide a high evidence level necessary to propose a classification and management algorithm.

Children with symptoms of unilateral or bilateral congenital nasolacrimal duct obstruction, no past surgical management, with one or more of the below criteria will be included:

1. Non-resolving symptoms of epiphora and/or discharge.
2. Congenital dacryocele not resolved after 1 week of lacrimal sac massage, and topical antibiotics.
3. As soon as subsidence of acute dacryocystitis. Parents will be asked about symptoms and patients will undergo lacrimal tests before and after operation in one week, one month and 3months based on a special record form. Patients will be randomly assigned to "simple probing" group or "endoscopy assisted probing" group.

All operations will be performed in operative theater and under general anesthesia. Pre- and post-operative examinations will be performed in plastic clinic in Farabi hospital.

DETAILED DESCRIPTION:
Congenital nasolacrimal duct obstruction is the most common cause of epiphora in infancy that can occur in 5% of newborn infants. It may resolve spontaneously in 95% of patients during the first year of life.(1) After that time surgical intervention is justified. Epiphora after birth is most commonly secondary to a developmental anomaly of imperforated membrane (Hasner valve) in distal part of nasolacrimal duct. Patients with congenital nasolacrimal duct obstruction (CNLDO) may show epiphora, eye discharge, acute dacryocystitis and cellulitis and dacryocele. Currently the management of primary CNLDO includes conservative treatment including lacrimal sac massage and topical antibiotics until 12 months of age.

The standard intervention for non-complicated, unresolved cases is simple blind probing of nasolacrimal duct. The overall success rate of one time simple probing is 75%-95 %. Simple probing is performed through a blind passage of a malleable metallic probe through punctum to nasolacrimal duct and inferior meatal space in nasal cavity.Although effective, probing may be associated with traumatic nasal bleeding, nasal mucosal damage,punctal and canalicular injury and false passage. The trauma is further concerned during stent insertion.In the past decade improvement in endoscopic instruments and techniques enabled us to visualize and smoothly manipulate anomalies in the nasal cavity and especially in the inferior meatus. Endoscopic assisted probing has been proposed as a measure to increase accuracy, efficacy and safety of nasolacrimal probing. Furthermore, by this method intranasal pathologies associated with failure of probing could be accurately diagnosed and specifically treated. To the best of our knowledge literature addressing this issue is limited to few limited case series.

The aim of this study is to compare results of endoscopy assisted nasolacrimal probing with the standard simple probing in cases with congenital nasolacrimal duct obstruction . Furthermore, investigators will identify associated anatomical anomalies. Investigators believe results of this study can be valuable in better understanding of this disease and provide a high evidence level necessary to propose a classification and management algorithm.

Children with symptoms of unilateral or bilateral congenital nasolacrimal duct obstruction, no past surgical management, with one or more of the below criteria will be included:

1. Non-resolving symptoms of epiphora and/or discharge.
2. Congenital dacryocele not resolved after 1 week of lacrimal sac massage, and topical antibiotics.
3. As soon as subsidence of acute dacryocystitis. Parents will be asked about symptoms and patients will undergo lacrimal tests before and after operation in one week, one month and 3months based on a special record form. Patients will be randomly assigned to "simple probing" group or "endoscopy assisted probing" group.

All operations will be performed in operative theater and under general anesthesia. Pre- and post-operative examinations will be performed in plastic clinic in Farabi hospital.

ELIGIBILITY:
Inclusion Criteria:

1. age: 3 weeks<Age<6 years
2. epiphora or discharge since birth or within 8 weeks after birth

Exclusion Criteria:

1. Follow up less than 3 months
2. Epiphora secondary to etiologies than congenital naso-lacrimal duct obstruction such as puncta/canalicular aplasia/dysgenesis;midfacial anomalies; congenital eyelid malposition;epiblepharon; trichiasis; congenital glaucoma, tumors; blepharitis; trauma Treatment success: defined success absence of epiphora/lacrimation and discharge 6 months after intervention.

Ages: 3 Weeks to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
success rate | 6 months
  absence of epiphora and discharge and negative dye disappearance test

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 month
  Incidence of complications related to the treatment including epistaxis, nasal stuffiness, injury to the nasolacrimal system or the eye, canalicular stenosis, keratopathy, nasal mucosa scar, synechia, tightening of inferior meatus (not reported at the time first intervention) to be described in those who need re-probing and nasal endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Farzad Pakdel, M.D., Principal Investigator — Farabi Hospital, Tehran University of Medical Sciences
Locations (1):
- Farzad Pakdel, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided